CLINICAL TRIAL: NCT01972100
Title: Use of Low-level Laser Therapy (808nm) to Muscle Fatigue Resistance: a Randomized Double-blind Crossover Trial
Brief Title: Use of Low-level Laser Therapy (808nm) to Muscle Fatigue Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleber Ferraresi (Other)
Collaborators: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Sponsor-Investigator, Cleber Ferraresi, Cleber Ferraresi, Universidade Federal de Sao Carlos
Organization: Universidade Federal de Sao Carlos (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP/UFRN 401/09
Record Dates: First submitted 2013-10-22; First posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Healthy
Keywords: Low-level laser therapy; Muscle fatigue resistance
MeSH Terms: interventions — Low-Level Light Therapy; Lasers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Low-level laser therapy (LLLT) (Active Comparator): Use of low-level laser therapy (LLLT) to induce a muscle fatigue resistance in intense exercises
  Interventions: Device: Low-level laser therapy (808nm); Other: isokinetic exercise
- Placebo low-level laser therapy (Placebo) (Active Comparator): Use of low-level laser therapy (LLLT) placebo to induce a muscle fatigue resistance
  Interventions: Other: isokinetic exercise; Device: Placebo low-level laser therapy

INTERVENTIONS:
Device: Low-level laser therapy (808nm) — Use of low-level laser therapy(LLLT)or placebo-LLLT applied on quadriceps femoris muscles between sets of isokinetic knee flexion-extension exercise
  Other Names: Low-level laser therapy;; Placebo low-level laser theraphy; Laser device (808nm; 100mW; DMC®, Brazil).
  Arms: Low-level laser therapy (LLLT)
Other: isokinetic exercise
  Other Names: Isokinetic knee flexion-extension exercise
Device: Placebo low-level laser therapy
  Arms: Placebo low-level laser therapy (Placebo)

SUMMARY:
The study hypothesis is a improved muscle fatigue resistance induced by low-level laser therapy applied between sets of intense exercises.

ELIGIBILITY:
Inclusion Criteria:

* healthy males
* physically active
* aged between 18-28 years old

Exclusion Criteria:

* smoker
* under medicine
* lower limb lesions limiting the flexion-extension of the knee joint

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Maximum repetitions | 1 week
  Evaluation of maximum repetitions of knee flexion-extension in isokinetic dynamometer. Volunteers were assessed on Monday (pre evaluation - baseline), on Wednesday performed a session of exercises and on Friday were assessed again (final evaluation).

SECONDARY OUTCOMES:
Median Frequency | 1 week
  Evaluation of median frequency by surface electromyography of quadriceps femoris muscles during maximum repetitions of knee flexion-extension in isokinetic dynamometer. Volunteers were assessed on Monday (pre evaluation - baseline), on Wednesday performed a session of exercises and on Friday were assessed again (final evaluation).

CONTACTS AND LOCATIONS:
Overall Officials: Cleber Ferraresi, MD, Principal Investigator — Universidade Federal de Sao Carlos; Wouber Hérickson de Brito Vieira, PhD, Study Director — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal Univesity of Rio Grande do Norte, Rio Grande Do Norte, Natal, Brazil

REFERENCES:
- [Background] Felismino AS, Costa EC, Aoki MS, Ferraresi C, de Araujo Moura Lemos TM, de Brito Vieira WH. Effect of low-level laser therapy (808 nm) on markers of muscle damage: a randomized double-blind placebo-controlled trial. Lasers Med Sci. 2014 May;29(3):933-8. doi: 10.1007/s10103-013-1430-2. Epub 2013 Sep 5. PMID 24005882
- [Background] Ferraresi C, Hamblin MR, Parizotto NA. Low-level laser (light) therapy (LLLT) on muscle tissue: performance, fatigue and repair benefited by the power of light. Photonics Lasers Med. 2012 Nov 1;1(4):267-286. doi: 10.1515/plm-2012-0032. PMID 23626925
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127
- [Background] Ferraresi C, de Brito Oliveira T, de Oliveira Zafalon L, de Menezes Reiff RB, Baldissera V, de Andrade Perez SE, Matheucci Junior E, Parizotto NA. Effects of low level laser therapy (808 nm) on physical strength training in humans. Lasers Med Sci. 2011 May;26(3):349-58. doi: 10.1007/s10103-010-0855-0. Epub 2010 Nov 18. PMID 21086010